CLINICAL TRIAL: NCT03481335
Title: Cluster Randomized Controlled Trial for a Community Health Promotion Program: Community Health Assessment Program in the Philippines (CHAP-P)
Brief Title: Community Health Assessment Program in the Philippines (CHAP-P)
Acronym: CHAP-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Ateneo de Zamboanga University (Other); Université de Montréal (Other); Global Alliance for Chronic Diseases (GACD) (Other); Canadian Institutes of Health Research (CIHR) (Other Government); International Development Research Centre, Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4303; 231837 (Other Grant/Funding Number: CIHR); 107826-001 (Other Grant/Funding Number: IDRC)
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Intervention Model Description: This study is a parallel 26-community cluster randomized controlled trial. A community cluster design was chosen as CHAP-P is intended as a community-level intervention. Thirteen communities (barangays) will receive the CHAP-P sessions and will be considered intervention, while the other 13 communities will receive care as usual and will be considered control. Measures of individual participants will be taken as a repeated cross-sectional sample at baseline and at six months. A community process evaluation and cost-effectiveness evaluation will also be undertaken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Community (Experimental): Intervention communities (barangays) will receive the intervention (CHAP-P sessions).
  Interventions: Other: CHAP-P Sessions
- Control Community (No Intervention): Control communities (barangays) will receive care as usual.

INTERVENTIONS:
Other: CHAP-P Sessions — Residents of intervention communities (barangays) aged 40+ are openly invited to attend CHAP-P sessions. At CHAP-P sessions, trained local volunteers (Barangay Health Workers, or BHWs) collect consent, measure blood pressure, collect other physical measurements, and conduct a survey to determine clients' risk of diabetes. Based on the findings, BHWs provide education and/or referrals. CHAP-P sessions are held twice a month, and clients are encouraged to continuing attending for ongoing follow-up and monitoring.
  Arms: Intervention Community

SUMMARY:
This study aims to evaluate the effectiveness of the Community Health Assessment Program in the Philippines (CHAP-P), looking at the differences between communities implementing CHAP-P versus communities not implementing CHAP-P.

DETAILED DESCRIPTION:
In this study, the investigators are evaluating the effectiveness of the CHAP-P intervention in communities of the Zamboanga Peninsula, Philippines. Specifically, the investigators are looking at the difference between hemoglobin A1c (HbA1c) levels in randomly selected residents of control communities versus those in communities implementing the CHAP-P intervention. The investigators are also looking at the differences between control and intervention communities in modifiable lifestyle risk factors for diabetes, screening rates for diabetes, rates of newly diagnosed cases of diabetes, general diabetes management, and hospital admission rates, as well as the cost effectiveness of CHAP-P.

The CHAP-P intervention consists of initial and follow-up sessions where trained local volunteers (Barangay Health Workers, or BHWs) take physical measurements (blood pressure, height, weight, waist circumference) and facilitate a diabetes risk survey; based on these findings, they provide education, materials, and referrals to local health resources as needed.

The participant groups in this evaluation include those that attend CHAP-P sessions, randomly selected community members that provide consent for a survey and HbA1c testing, and community members and BHWs/other Lead Local Organization staff who provide consent for focus groups and interviews.

ELIGIBILITY:
Inclusion Criteria (Community Survey Participants & CHAP-P Session Participants):

* Aged 40 years of age or older
* Resident of community

Exclusion Criteria (Community Survey Participants & CHAP-P Session Participants):

* Under 40 years of age
* Resident of a different community

Inclusion Criteria (Barangay Health Workers [BHW]/Lead Local Organization [LLO] Staff)

- Must be a BHW or other LLO staff who is participating in the CHAP-P Intervention

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5229 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline, 6 months
  Mean difference in HbA1c at 6 months in the intervention group compared to the control group. Measured with the A1CNow+ point-of-care device in a community location after the completion of the in-home community survey.

SECONDARY OUTCOMES:
Physical Activity | Baseline, 6 months
  Mean difference in physical activity at 6 months in the intervention group compared to the control group. Measured with the International Physical Activity Questionnaire (International Physical Activity Quotient, IPAQ), included in the community survey.
Medication Compliance | Baseline, 6 months
  Mean difference in medication compliance at 6 months in the intervention group compared to the control group. Self-reported, via community survey questions.
Blood Pressure | Baseline, 6 months
  Mean difference in blood pressure at 6 months in the intervention group compared to the control group. Measured using a blood pressure device, the Microlife WatchBP Office Target.
Community Residents Newly Diagnosed with Diabetes | 6 months
  Mean difference in number of community residents newly diagnosed with diabetes at 6 months in the intervention group compared to the control group. Numbers taken from Rural Health Unit databases
Hospital admission rates | -12 months, 12 months
  Mean difference in hospital admission rates due to diabetes and diabetes-related conditions, hypertension, myocardial infarction, stroke, congestive heart failure at 6 months in the intervention group compared to the control group. Numbers taken from central Department of Health database (12 months before and 12 month after CHAP-P implementation, and divided by mid-year population estimates)
Mortality rates | -12 months, 12 months
  Mean difference in mortality rates due to diabetes and diabetes-related conditions, hypertension, myocardial infarction, stroke, congestive heart failure based on International Classification of Disease (ICD)-10 codes at 6 months in the intervention group compared to the control group. Numbers taken from Regional Field Health Surveillance Information Systems (measured 12 months before and 12 month after CHAP-P implementation, 6 month estimated by dividing by mid-year population estimates)
Quality of Life (EQ5D-5L) | Baseline, 6 months
  Mean difference in quality of life at 6 months in the intervention group compared to the control group. Measured with the EuroQol-5 dimension-5 level (EQ5D-5L), included in the community survey
Knowledge about Diabetes and Hypertension | Baseline, 6 Months
  Mean difference in knowledge about diabetes and hypertension at 6 months in the intervention group compared to the control group. Measured with elements of the Health Awareness and Behaviour Tool (HABiT) included in the community survey.
Risk Factors for Diabetes | Baseline, 6 months
  Mean difference in risk factors for diabetes at 6 months in the intervention group compared to the control group. Measured with the Finnish Diabetes Risk Score (FINDRISC), included in the community survey
Risk Behaviours for Diabetes/Cardiovascular Issues | Baseline, 6 months
  Mean difference in risk behavhiours for diabetes/cardiovascular issues (activity, diet, smoking, alcohol, stress) at 6 months in the intervention group compared to the control group. Measured with elements of the Health Awareness and Behaviour Tool (HABiT) included in the community survey.
Perceived Concern and Understanding of Risk | Baseline, 6 months
  Mean difference in perceived concern and understanding of risk at 6 months in the intervention group compared to the control group. Measured with elements of the Health Awareness and Behaviour Tool (HABiT) included in the community survey.
Confidence in Behaviour Change | Baseline, 6 months
  Mean difference in confidence in behaviour change at 6 months in the intervention group compared to the control group. Measured with elements of the Health Awareness and Behaviour Tool (HABiT) included in the community survey.
Quality-Adjusted Life Years (QALYs) | 12 months
  Secondary; calculated from the EQ5D-5L.
Cost-effectiveness | 12 months
  Comparing program cost of implementing CHAP-P (collected via team tracking) and healthcare resource utilization costs (collected via self-report from participants during community survey) to percentage reduction in HbA1c and blood pressure.
Cost-utility | 12 months
  Cost of program and healthcare resource utilization costs per QALY

CONTACTS AND LOCATIONS:
Overall Officials: Gina Agarwal, MBBS, PhD, Principal Investigator — McMaster University; Fortunato Cristobal, MD, MPH, MHPEd, Principal Investigator — Ateneo de Zamboanga University
Locations (1):
- Ateneo de Zamboanga University, Zamboanga City, Zamboanga Del Sur, Philippines

REFERENCES:
- [Derived] Agarwal G, Angeles RN, Dolovich L, Kaczorowski J, Gaber J, Guenter D, Arnuco FD, Lam HY, Thabane L, O'Reilly D, Agbulos RM, Arciaga RS, Barrera J, Gregorio E, Halili S Jr, Jalani N, Cristobal F. The Community Health Assessment Program in the Philippines (CHAP-P) diabetes health promotion program for low- to middle-income countries: study protocol for a cluster randomized controlled trial. BMC Public Health. 2019 Jun 3;19(1):682. doi: 10.1186/s12889-019-6974-z. PMID 31159778